| Consent Form, | 1 <sup>st</sup> July 2017. | Version 1 |
|---------------|----------------------------|-----------|

## Sleep, Wake and Light therapy for depression

**Informed Consent Form** 

1st July 2017



Ethics Approval Reference: 17/LO/1567, IRAS Project ID: 225748

## **CONSENT FORM**

Title of Project: Sleep, Wake and Light therapy for depression

Name of Researcher: Professor David Veale

Please initial the boxes

researchers.

| 1. | I confirm that I have read the information sheet dated 1 <sup>st</sup> July 2017 (version 1) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals attached to the research study, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared <i>anonymously</i> with other |

| Cons | ent Form, 1 <sup>st</sup> July 2017, | Version 1 | |
|---|---|---|---|
| 5. | , | eneral Practitioner being informed of my participation in the any necessary exchange of information about me between my arch team. | |
| 6. | I agree to take part ir | n the above study. | |
| Nam | e of Participant | Date | Signature |
| Nam | ne of Person | <br>Date | Signature |

taking consent